CLINICAL TRIAL: NCT00776880
Title: Reevaluating the American Society of Anesthesiologists (ASA) Physical Status System in Patients Assessment and Compared With a New Scale of Physical-psycho-social Gauge Raised by Our Institution
Brief Title: Does American Society of Anesthesiologists (ASA) Physical Status Scale Enough in Patients Assessment
Acronym: ASAINPA
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Other Study IDs: NMU-FY2008-MZ08; NJFY080921
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-11

CONDITIONS: Elective Surgery
Keywords: Surgical operation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients assessed with ASA physical status scale
  Interventions: Other: ASA scale
- 2: Patients assessed with PPS scale
  Interventions: Other: PPS scale

INTERVENTIONS:
Other: ASA scale — ASA scale evaluation before operation
  Groups: 1
Other: PPS scale — PPS scale evaluation before operation
  Groups: 2

SUMMARY:
American Society of Anesthesiologists (ASA) physical status scale has been used worldwide for assessing the status of patients before operation. However, merely the value of ASA scale did not give enough information of patients to determine their prognosis and improvement of outcomes. Since 1948, World Health Organization (WHO) defined health as the state of complete physical, mental and social well-being and not merely the absence of disease or infirmity. Therefore, the investigators hypothesized that the ASA scale only was needed to be modified and should be replaced by a comprehensive gauge to evaluate the status of patients in depth. Based on this thought, the investigators used a new system, i.e., physical-psycho-social (PPS) scale, to assess the overall state before surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgical operation
* Age from 18-65 years

Exclusion Criteria:

* Age < 18 years or > 65 years
* Not willing to participate in this study
* Patients from emergency department

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgical operations
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time of recovery | Six months after operation.

SECONDARY OUTCOMES:
Intraoperative consumption of drugs | 1 day after operation
Incidence of side events | 72 hours after operation
Hospitalization days | From 0 min after operation to the time duration of discharge home, this measure would be varied in different patients
Psychological state | Six months after operation
Life quality | Six months after operation

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China